CLINICAL TRIAL: NCT05488600
Title: Comparison of the Executive Functions of Elite Team-Sport and Individual-Sport Athletes
Brief Title: Executive Functions in Elite Athletes
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mehmet akif akinci, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: AkifAkinci
Record Dates: First submitted 2022-07-13; First posted 2022-08-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Cognitive Change
Keywords: Elite Athletes; Executive Function; Cognition; Sports; Team Sports
MeSH Terms: interventions — Neuropsychological Tests; Stroop Test; Trail Making Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Team Sports: 30 elite athletes between the ages of 20-30 who are interested in team sports
  Interventions: Behavioral: Executive Function Assessment
- Individual Sports: 30 elite athletes between the ages of 20-30 who are interested in individual sports
  Interventions: Behavioral: Executive Function Assessment
- Control Group: 30 healthy individuals between the ages of 20-30 who are not interested in sports
  Interventions: Behavioral: Executive Function Assessment

INTERVENTIONS:
Behavioral: Executive Function Assessment — Digit Span (Forward and Backward) Test, Stroop Test, Trail Making Test A and B forms, Tower of London Test were used to evaluate executive functions.
  Other Names: Digit Span Test; Stroop Test; Trail Making Test; London Tower Test

SUMMARY:
In the study, it was aimed to compare the executive functions of elite athletes who do team sports and individual sports with each other and with individuals who do not do sports.

DETAILED DESCRIPTION:
In the study, it was aimed to compare the executive functions of elite athletes who do team sports and individual sports with each other and with individuals who do not do sports. 60 elite athletes participating in national and international competitions between the ages of 20-30, affiliated to the Republic of Turkey Ministry of Youth and Sports and federations, and 30 individuals who did not do sports for the control group were included in the study group. Of the elite athletes, 30 were included in the team sports group and 30 in the individual sports group. Executive functions Forward and Backward Digit Span Test, Stroop Test, Trail Making Test A and B form (TMT-A, TMT-B) and Tower of London (ToL) Test evaluated with.

ELIGIBILITY:
Inclusion Criteria:

* Be between 20-30 years old
* Have been doing sports for at least 5 years
* Being an elite athlete
* Being actively involved in sports

Exclusion Criteria:

* Having any psychological or neurological disease

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elite athletes participating in national and international competitions in Turkish Basketball Federation, Turkish Volleyball Federation and Turkish Football Federation clubs and Gaziantep Youth Sports Center
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
London Tower Test | day 1
  The Tower of London test is an executive function test that is particularly sensitive to planning and problem-solving skills. The Tower of London test consists of 2 tower boards and red, blue and green beads. The participant is asked to make the same shape on the tower board of the tester opposite him on his own tower board in the fewest moves. A low total score and a high correct total score indicate good planning and problem-solving abilities. The high score of total rule mistake indicates the negativities in the ability to acquire and control planning and problem-solving behavior under certain rules. The excess of the total time out indicates the difficulty in planning and problem-solving skills at a certain time. The shortness of the onset time indicates effective planning before the problem-solving response begins. The application time and the shortness of the total time indicate the speed of problem-solving.

SECONDARY OUTCOMES:
Digit Span Test | day 1
  The test consists of two parts forward and backward span. The participant is asked to repeat the numbers read in one second intervals in the forward span in the same order. It assesses attention, concentration and short-term memory. In the backward span, the numbers read at one-second intervals are requested to be repeated in reverse order from the end to the beginning. Working memory, which is a component of executive functions, is evaluated. The highest score that can be obtained for the forward span is 8 points, and 7 for the backward span, for a total of 15 points.
Stroop Test | day 1
  The Stroop test evaluates inhibitory control, which is a component of executive functions. On the card we used as test material, the words blue, green, red, yellow are written and painted in a different color than the word. The person is first asked to read the colored words printed unrelated to the color. In the second step, the person is asked to say the color of the colored words written unrelated to the color on which they are printed. The time from the "start" command to the end, the number of errors and corrections are recorded. The time difference between the two stages constitutes the interference score. Error and correction numbers are calculated. The long duration of interference, errors and corrections indicate that the person's attention is easily distracted and cannot suppress inappropriate stimuli.
Trail Making Test | day 1
  The Trail Making test consists of two parts, A and B. In part A, the participants are asked to combine the circles with numbers randomly scattered on the paper in the correct order and follow each other (1-2-3-4-5...). In section B, there are letters and numbers randomly placed in circles. Participants are asked to combine a letter and a number in the correct sequence (1-A-2-B-3-C-4-D...) consecutively. Time is kept for both sections. The duration is expected to be short. The A part of the TMT evaluates the processing speed based on visual scanning ability, and the B part evaluates the complex attention, planning, set changing, inhibition ability, and following the sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Meng FW, Yao ZF, Chang EC, Chen YL. Team sport expertise shows superior stimulus-driven visual attention and motor inhibition. PLoS One. 2019 May 15;14(5):e0217056. doi: 10.1371/journal.pone.0217056. eCollection 2019. PMID 31091297
- [Result] De Waelle S, Laureys F, Lenoir M, Bennett SJ, Deconinck FJA. Children Involved in Team Sports Show Superior Executive Function Compared to Their Peers Involved in Self-Paced Sports. Children (Basel). 2021 Mar 30;8(4):264. doi: 10.3390/children8040264. PMID 33808250